CLINICAL TRIAL: NCT01985646
Title: A Prospective, Randomized Controlled Trial of Conservative Versus Surgery Treatment of Normal and Short-segment Hirschsprung Disease for Infants
Brief Title: A Trial on Conservative Treatment for Infants' Hirschsprung Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jiexiong Feng, professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001; 20090302 (Other: TongjiHospital)
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung disease; conservative treatment; surgery treatment; infants
MeSH Terms: conditions — Hirschsprung Disease | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery treatment (Experimental): one stage pull through left-colectomy
  Interventions: Procedure: surgery treatment
- conservative treatment (Experimental): anal dilation, colonic lavage, oral probiotic
  Interventions: Behavioral: anal dilation; Behavioral: colonic lavage; Drug: oral probiotic

INTERVENTIONS:
Procedure: surgery treatment — one staged pull-through left-colectomy
  Arms: surgery treatment
Behavioral: anal dilation — anal dilation
  Arms: conservative treatment
Behavioral: colonic lavage — colonic lavage
  Arms: conservative treatment
Drug: oral probiotic — oral probiotic
  Arms: conservative treatment

SUMMARY:
The present study was designed to compare the efficacy of conservative treatment to operative treatment for improvement of constipation symptoms in infants with short or normal-segment Hirschsprung disease.

ELIGIBILITY:
Inclusion Criteria:

* Hard or firm stools for twice or less per week
* Age were from newborn to 3 months
* Histochemical acetylcholinesterase reaction (AChE) in rectal mucosa was positive
* The narrowed distal bowel on barium enema was characterized as normal or short-segment Hirschsprung disease with a 24h barium retention

Exclusion Criteria:

* Children >3months of age
* Patients presented severe inflammation or malnutrition, unconsciousness, and symptoms of a ruptured hollow viscus
* Barium enema showed long-segment or total colonic aganglionic bowel

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
the change of defecation frequence | 6~12 months
  the changes of defecation frequence at 6~12 months after treatment

SECONDARY OUTCOMES:
stool pattern | 6~12 months
  stool pattern as Forming soft stool or Loose stool
controlling defecation ability | 6~12 months
  whether patients' controlling of defecation be better or not after treatment
complications | 6~12 months
  complications were suffered by patients or not, such as enterolitis, anastomotic stenosis etc.